CLINICAL TRIAL: NCT02966743
Title: Effect of Medazolam or Dexmedetomidine on Regional Cerebral Oxygen Saturation During Spinal Anesthesia in the Elderly Patients
Brief Title: Effect of Sedatives on Regional Cerebral Oxygen Saturation
Acronym: 2
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Youn Yi Jo, Assistant professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GCIRB2016-293
Record Dates: First submitted 2016-11-08; First posted 2016-11-17 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Cerebral Ischemia-Hypoxia
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Midazolam; Dexmedetomidine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- midazolam (Experimental): administration of midazolam during spinal anesthesia for target bispectral index 75-80
  Interventions: Drug: Midazolam
- dexmedetomidine (Active Comparator): administration of dexmedeomidine during spinal anesthesia for target bispectral index 75-80
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Midazolam — administration of midazolam during spinal anesthesia for target bispectral index 75-80
  Other Names: Mida
  Arms: midazolam
Drug: Dexmedetomidine — administration of dexmedetomidine during spinal anesthesia for target bispectral index 75-80
  Other Names: Dex
  Arms: dexmedetomidine

SUMMARY:
Compare the changes of regional cerebral oxygen saturation during midazolam or dexmedetomidine sedation for spinal anesthesia in the elderly patients who undergoing femur surgery.

DETAILED DESCRIPTION:
Compare the changes of regional cerebral oxygen saturation during midazolam or dexmedetomidine administration (target bispectrl index 75-80) for spinal anesthesia in the elderly patients over 65 years who undergoing femur surgery.

ELIGIBILITY:
Inclusion Criteria:

* patinets who undergoing femur surgery under spinal anesthesia

Exclusion Criteria:

* previous cerebrovascular disease, uncontrolled cardiovascular disorder, uncontrolled pulmonary disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
regional cerebral oxygen saturation | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Youn Yi Jo, MD, Study Director — Gachon University Gil Medical Center
Locations (1):
- Gachon University Gil Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: Undecided